CLINICAL TRIAL: NCT06432374
Title: Open Pilot of Written Exposure Therapy for Nurses Experiencing Work-Related Posttraumatic Stress
Brief Title: Written Exposure Therapy for Nurses
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Yang Li, Assistant Professor, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00203166
Record Dates: First submitted 2024-05-21; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Posttraumatic Stress Disorder; Depressive Symptoms; Burn Out; Anxiety; Work Related Stress
Keywords: Nurses; Written Exposure Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Burnout, Psychological; Anxiety Disorders; Occupational Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Written Exposure Therapy (Experimental): WET is a trauma-focused therapy for PTSD. It includes five writing sessions.
  Interventions: Behavioral: WET

INTERVENTIONS:
Behavioral: WET — The five weekly WET sessions were delivered online via Canvas. Five session modules were created, each containing writing instructions for the respective session and an assignment feature for participants to upload their narratives. All sessions included 30 minutes of writing. Following instructions, participants wrote about a specific work-related trauma event in detail and described the emotions and thoughts experienced during the event. While all sessions were self-paced, participants were advised to complete each subsequent session within one week. Participants had the option to self-administer sessions or participate in Zoom "office hours" for live writing sessions with a facilitator who had completed WET training providing the writing instructions.

SUMMARY:
Nurses often experience elevated levels of stress, overwork, and trauma in the workplace, leading to posttraumatic stress disorder (PTSD), depression, burnout, and even nurse turnover. While effective therapies for PTSD exist, barriers to treatment arise from nursing culture, such as workplace stigma about mental health problems, fear that psychological status may impact performance evaluations, and demands of shiftwork. There is a pressing need for scalable evidence-based interventions tailored to nursing culture to effectively address PTSD and related mental health issues. The study aimed to assess the feasibility, safety, and acceptability of a tailored evidence-based treatment, Written Exposure Therapy (WET), for nurses experiencing work-related traumatic stress.

This single-arm open pilot study with pre- and post-intervention assessments, included participants from two nursing schools' alumni. Eligibility criteria included nurses screening positive for work-related trauma with a report of at least two PTSD symptoms. Participants engaged in a self-administered, asynchronous, five-week online writing session, facilitated by WET-trained nurses. Outcomes measures (PTSD, depression, anxiety, burnout, and intention to quit) were assessed at baseline, post-intervention, and 5-weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Work-related trauma
* Posttraumatic stress disorder

Exclusion Criteria:

* Current substance abuse
* Current suicidality
* Current psychiatric treatment with psychotherapy or psychotropic medications other than selective serotonin (and norepinephrine) reuptake inhibitors (SSRI/SNRI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Posttraumatic stress disorder | Baseline, immediately post-intervention, and 5 weeks follow-up
  The PTSD Checklist for DSM-5 was used to assess symptoms of posttraumatic stress disorder in the past month. The total score ranges from 0-80, with higher scores indicating more severe PTSD symptoms.

SECONDARY OUTCOMES:
Depression | Baseline, immediately post-intervention, and 5 weeks follow-up
  The Patient Health Questionnaire-8 was used to assess the frequency of depressed mood in the past two weeks. The total score ranges from 0-24, with higher scores indicating more severe depression symptoms.
Anxiety | Baseline, immediately post-intervention, and 5 weeks follow-up
  The Generalized Anxiety Disorder-7 was used to assess the frequency of anxiety symptoms in the past two weeks. The total score ranges from 0-21, with higher scores indicating more severe anxiety symptoms.
Professional Quality of Life | Baseline, immediately post-intervention, and 5 weeks follow-up
  The Professional Quality of Life was used to assess compassion satisfaction, burnout, and secondary traumatic stress. Each subscale score ranges from 10-50, with higher scores indicating higher levels of compassion satisfaction, more burnout symptoms, and more secondary traumatic stress.
Intention to Quit | Baseline, immediately post-intervention, and 5 weeks follow-up
  Intention to quit the job or leave the nursing profession were asked using two questions - "How often have you thought about quitting your job in the past month?", "How often have you thought about leaving the nursing profession in the past month?". The five responses are "never," "rarely," "sometimes," "very often", and "always." The scores for both intention to quit the job and intention to leave the nursing profession range from 1-5, with higher scores indicating greater intention to quit the job or leave the nursing profession.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States